CLINICAL TRIAL: NCT02206360
Title: Observational Study to Analyze the Outcomes of Subjects Who - Based Upon Their Sufficiently Elevated Risk for the Development of Pancreatic Adenocarcinoma- Elect to Undergo Early Detection Testing
Brief Title: Pancreatic Cancer Early Detection Program
Acronym: PCEDP
Status: Active, not recruiting | Type: Observational
Sponsor: White Plains Hospital (Other)
Responsible Party: Principal Investigator, Joshua Raff, MD, Director, Digestive Cancer Program, Center for Cancer Care, White Plains Hospital
Other Study IDs: WPH 1401
Record Dates: First submitted 2014-07-29; First posted 2014-08-01 (Estimated); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Pancreatic Cancer; Pancreas Cancer; Pancreatic Adenocarcinoma; Familial Pancreatic Cancer; BRCA 1/2; HNPCC; Lynch Syndrome; Hereditary Pancreatitis; FAMMM; Familial Atypical Multiple Mole Melanoma; Peutz Jeghers Syndrome
Keywords: Pancreatic Cancer; Pancreatic Cancer Screening; Pancreas Cancer; Pancreatic Adenocarcinoma; Pancreatic Adenocarcinoma screening; Familial Pancreatic Cancer; BRCA 1/2; HNPCC; Lynch Syndrome; Hereditary Pancreatitis; FAMMM; Familial atypical multiple mole melanoma; Peutz Jeghers Syndrome; MRI; Magnetic Resonance Imaging; EUS; Endoscopic Ultrasound; Early detection; Screening
MeSH Terms: conditions — Pancreatic Neoplasms; Pancreatic carcinoma, familial; Colorectal Neoplasms, Hereditary Nonpolyposis; Hereditary pancreatitis; Dysplastic Nevus Syndrome; Peutz-Jeghers Syndrome | interventions — Endoscopic Ultrasound-Guided Fine Needle Aspiration; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Individuals at elevated risk for pancreatic cancer: Individuals with an elevated risk of developing pancreatic cancer as either equal to or greater than five times the general population risk, or five times the average risk (1.5%) of developing pancreatic cancer by age 70; that is a 7.5% lifetime risk.
  Interventions: Procedure: Endoscopic Ultrasound; Procedure: Magnetic Resonance Imaging (MRI)

INTERVENTIONS:
Procedure: Endoscopic Ultrasound
Procedure: Magnetic Resonance Imaging (MRI)

SUMMARY:
Early detection testing is recommended for individuals at elevated risk for the development of Pancreatic Cancer. This Protocol will define sufficiently elevated risk as either equal to or greater than five times the general population risk, or five times the average risk (1.5%) of developing pancreatic cancer by age 70; that is a 7.5% lifetime risk. Our inclusion criteria has a strong focus on the risk for pancreatic cancer imparted by the presence of hereditary cancer genes, as well as by family history. Enrolled subjects will undergo Endoscopic Ultrasound (EUS) alternating with Magnetic Resonance Imaging (MRI), every six to 12 months, for up to 5 years.

DETAILED DESCRIPTION:
Interested individuals can be referred by physicians, or by family or friends.

Individuals are informed that the purpose of this study is to collect outcome data following early detection testing based upon our criteria for elevated risk.

Consent is obtained by any of the co-investigators. Consent is obtained for the primary PCEDP, and also obtained to allow for data to be used by our Cancer Program.

We have a weekly review of all calls made and of all enrollments.

We have a monthly meeting to review all proceeding regarding the study.

Our IRB routinely reviews the proceedings of the study

Our institution has a monthly Clinical research Committee meeting.

ELIGIBILITY:
Inclusion Criteria: Any of the following:

1. Known carrier of either the BRCA2 or CDKN2A mutation;
2. Known carrier of any of the following mutations (BRCA1, MLH1, MSH2, PMS2, MSH6, EPCAM , P53, PALB2, APC, or ATM) PLUS first or second degree relative affected with pancreatic cancer;
3. Individual with Peutz-Jeghers Syndrome;
4. Familial Pancreatic Cancer, defined as at least two affected relatives with Pancreatic Cancer, who are first degree relatives with each other, and at least one of those affected must be first degree relative to the study subject;
5. Both parents affected, any age:
6. Any first degree relative diagnosed with pancreatic cancer under age 50;
7. Chronic Pancreatitis Syndrome, defined by either PRSS1 or SPINK1 mutations AND appropriate clinical and family history

Exclusion Criteria:

1. Any medical condition that contraindicates endoscopy or biopsy
2. Any medical condition that contraindicates MRI
3. Status post partial or complete resection of the pancreas
4. History of pancreatic cancer, either endocrine or exocrine
5. Clinical suspicion of pancreatic cancer, or any previous radiographic or histologic diagnosis of a pre-malignant finding, including IPMN (Intraductal papillary mucinous neoplasm) and PanIN (Pancreatic intraepithelial Neoplasm).
6. diagnosis of dementia
7. Uncontrolled, current illness
8. Renal insufficiency with serum creatinine greater than 2.0 mg/dl

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals aged 18 and older, who carry sufficiently elevated risk for the development of pancreatic cancer, numerically defined as over (or near) 5 times the general population risk, as determined by their personal, familial, or genetic history.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2014-04; Primary Completion 2024-03 (Actual); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Premalignant or malignant pancreatic conditions found with alternating EUS and MRI testing. | 5 years
  Number of Participants with Premalignant or Malignant Pancreatic Conditions, as a Measure of Safety and Efficacy

SECONDARY OUTCOMES:
Clinical outcomes which occur as a result of this Protocol | 5 years
  Prospective collection and reporting of any malignant conditions which occur as a result of this Protocol, including from surgery, or other testing.
Complications of any interventions as a result of this Protocol | 5 years
  Prospective collection and reporting of any complications that may be associated with early detection testing, including hospitalization, disability, and death.
Non-Pancreatic cancers diagnosed while on this protocol | 5 years
  Prospective collection and reporting of non-pancreatic cancers detected during this Protocol, including pancreatic cysts.

CONTACTS AND LOCATIONS:
Locations (1):
- White Plains Hospital, White Plains, New York, United States

REFERENCES:
- [Derived] Raff JP, Cook B, Jafri FN, Boxer N, Maldonado J, Hopkins U, Roayaie S, Noyer C. Successful Pancreatic Cancer Screening Among Individuals at Elevated Risk Using Endoscopic Ultrasound and Magnetic Resonance Imaging: A Community Hospital Experience. Pancreas. 2022 Nov-Dec 01;51(10):1345-1351. doi: 10.1097/MPA.0000000000002182. PMID 37099777